CLINICAL TRIAL: NCT01877408
Title: A Randomized Controlled Trial of Open Surgical vs. Rapid, Minimally-invasive Voluntary Adult Male Circumcision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Simunye Primary Health Care (Other)
Responsible Party: Principal Investigator, Peter Millard, PI, Simunye Primary Health Care
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNICIRC SA
Record Dates: First submitted 2013-06-11; First posted 2013-06-13 (Estimated); Results first posted 2014-02-06 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Circumcision
Keywords: disposable circumcision device; Tissue adhesive; Open surgical circumcision; Minimally-invasive circumcision
MeSH Terms: interventions — Tissue Adhesives

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open surgical circumcision (Active Comparator): The open surgical technique, which is commonly used for circumcision in South Africa, requires good surgical skills and minor complications are common.
  Interventions: Procedure: Open surgical circumcision
- Unicirc device with tissue adhesive (Experimental): Coupling removal of the foreskin using the disposable Unicirc device with wound sealing using tissue adhesive results in a procedure that can be performed by generalist doctors with minimal training.
  Interventions: Device: Unicirc device with tissue adhesive

INTERVENTIONS:
Procedure: Open surgical circumcision — Open surgical circumcision using a technique approved by the WHO (dorsal slit)
  Arms: Open surgical circumcision
Device: Unicirc device with tissue adhesive — Removal of foreskin with Unicirc disposal device and wound sealing with tissue adhesive.
  Arms: Unicirc device with tissue adhesive

SUMMARY:
To identify a minimally-invasive surgical circumcision technique for men, which is easy to learn and perform, is safe, and is associated with high patient satisfaction and excellent cosmetic results.

DETAILED DESCRIPTION:
Voluntary medical male circumcision (VMMC) is a priority preventive intervention for HIV transmission. Currently, the most widely used VMMC technique in South Africa is open surgical circumcision.

According to the Framework for Clinical Evaluation of Devices for Adult Male Circumcision (WHO, 2011): "WHO and other health authorities wish to identify one or more devices that (a) would make the VMMC safer, easier, and quicker; (b) would have more rapid healing than current methods and/or might entail less risk of HIV transmission in the post-operative period; (c) could be performed safely by health-care providers with a minimal level of training; and (d) would be cost-effective compared to standard surgical methods for male circumcision scale up."

This randomized controlled trial compares the open surgical technique to an alternative minimally-invasive technique using a disposable Unicirc device with tissue adhesive. The investigators postulate that VMMC using the Unicirc device meets WHO criteria for the ideal method to scale up: it is an easier technique to learn and perform, requires less intraoperative time, is safer for both surgeons and patients, heals quicker, and is more cost effective than other currently available techniques. The disposable nature of the device is an immense advantage as it eliminates the need to sterilize and can therefore be used in resource-limited settings. It also reduces the chances of infection caused by contaminated instruments.

The study will randomly assign participants to one of two groups:

* Unicirc device with tissue adhesive: 100 men
* Open surgical circumcision: 50 men

The participants will be evaluated during follow-up visits at 2 days, 7 days, 14 days, and 28 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men at least 18 years of age requesting circumcision
* No anatomical penile abnormalities or infections
* Able to provide informed consent to participate
* Willing to participate in follow-up visits

Exclusion Criteria:

* Current illness
* Penile abnormality or infection which contraindicates or would complicate circumcision
* History of bleeding disorder
* Past reaction to local anesthetic

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Millard, MD, PhD, Principal Investigator — Simunye Primary Health Care
Locations (1):
- Simunye Primary Healthcare, Mitchells Plain, Western Cape, South Africa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between 31 May, 2013 and 26 June, 2013. Participants were recruited via posters at two affiliated primary care clinics in Cape Town.
Pre-assignment Details: Healthy, uncircumcised men who were at least 18 years of age were eligible to participate in the study. All those who were enrolled and who showed up for their procedure were included in the study.
Period: Overall Study
Arm/Group | Open Surgical Circumcision | Unicirc Device With Tissue Adhesive
Started | 50 | 100
Completed | 50 (Completed follow up visit 28 days after procedure) | 98 (Completed follow up visit 28 days after procedure)
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Open Surgical Circumcision | Unicirc Device With Tissue Adhesive | Total
Number analyzed (Participants) | 50 | 100 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 100 | 149
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 50 | 100 | 150
Region of Enrollment [Number; unit: participants]
  South Africa | 50 | 100 | 150

OUTCOME MEASURES:

1. Primary Outcome: Intraoperative Duration
Description: Amount of time from first manipulation of tissue under local anesthesia to dressing
Time Frame: 1 hour
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Open Surgical Circumcision | Unicirc Device With Tissue Adhesive
Number analyzed (Participants) | 50 | 100
minutes
  Procedure without frenulectomy (n=44,96) | 22.6 (8.6) [14 to 31.2] | 13.0 (4.5) [8.5 to 17.5]
  Procedure with frenulectomy (n=6,4) | 25.0 [7 to 43] | 28.6 [10.9 to 46.3]

2. Secondary Outcome: Difficulty in Learning and Performing Technique
Description: Evaluated by doctor survey based on 5 point Likert scale
  1. Unicirc is much easier
  2. Unicirc is easier
  3. Neutral
  4. Open surgical is easier
  5. Open surgical is much easier
Time Frame: 1 year
Population: The four physicians that participated in this study performed both procedures (i.e. open surgical and Unicirc) on study participants. Three physicians had significant previous (non-study) experience performing open surgical circumcisions. All four had no to very limited previous experience performing Unicirc circumcisions.
Measure: Median (Full Range); unit: units on Likert scale
Groups:
- Physicians: The generalist doctors in this study were moderately experienced in open surgical circumcision but had not previously used the Unicirc instruments.
Arm/Group | Physicians
Number analyzed (Participants) | 4
units on Likert scale | 2 [1 to 5]

3. Secondary Outcome: Number of Participants With Complete Wound Healing by Post-Surgery Week 4
Time Frame: Within 4 weeks after surgery
Measure: Number; unit: participants
Arm/Group | Open Surgical Circumcision | Unicirc Device With Tissue Adhesive
Number analyzed (Participants) | 50 | 98
participants | 49 | 89

4. Secondary Outcome: Pain Experienced
Description: Pain experienced during and after the procedure evaluated using a 10 point pain scale (0 signifies no pain and 10 signifies maximal pain
Time Frame: Within 2 days after surgery
Measure: Mean (Standard Deviation); unit: units on a 10-point pain scale
Arm/Group | Open Surgical Circumcision | Unicirc Device With Tissue Adhesive
Number analyzed (Participants) | 50 | 100
units on a 10-point pain scale
  Pain in first 24 hours post-op | 3.1 (2.4) | 4.2 (2.7)
  Pain at 48 hours post-op | 1.2 (2.0) | 0.7 (1.6)

5. Secondary Outcome: Overall Patient Satisfaction
Description: Patient satisfaction evaluated with questionnaire using satisfaction scale
  1. Very satisfied
  2. Satisfied
  3. Not satisfied
Time Frame: Within 6 weeks after surgery
Measure: Number; unit: participants
Arm/Group | Open Surgical Circumcision | Unicirc Device With Tissue Adhesive
Number analyzed (Participants) | 50 | 98
participants
  Very satisfied | 40 | 78
  Satisfied | 8 | 15
  Not satisfied | 2 | 5

6. Secondary Outcome: Cosmetic Result
Description: Cosmetic result evaluated by classification of scar line as regular (straight without any irregularity), irregular (not completely straight), or scalloped (with a wavy appearance)
Time Frame: Within 6 weeks after surgery
Measure: Number; unit: participants
Arm/Group | Open Surgical Circumcision | Unicirc Device With Tissue Adhesive
Number analyzed (Participants) | 50 | 98
participants
  Regular | 20 | 79
  Irregular | 8 | 12
  Scalloped | 22 | 7

7. Other Pre Specified Outcome: Number of Participants With Adverse Events
Description: Number of participants with intraoperative and post-operative adverse events, such as bleeding, hematoma, and infection
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Open Surgical Circumcision | Unicirc Device With Tissue Adhesive
Number analyzed (Participants) | 50 | 100
participants
  Mild bleeding | 1 | 4
  Moderate bleeding (suturing required) | 2 | 10
  Hematoma | 0 | 4
  Infection (antibiotic required) | 6 | 10

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Open Surgical Circumcision | Unicirc Device With Tissue Adhesive
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/100
Other Adverse Events (participants affected / at risk) | 9/50 | 28/100
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Surgical Circumcision (N=50) | Unicirc Device With Tissue Adhesive (N=100)
Mild post-operative bleeding (Surgical and medical procedures) | 1 (1) | 4 (4)
Moderate post-operative bleeding (Surgical and medical procedures) | 2 (2) | 10 (10) — Required suturing to stop bleeding
Hematoma (Surgical and medical procedures) | 0 (0) | 4 (4)
Post-operative infection (Surgical and medical procedures) | 6 (6) | 10 (10) — Required antibiotic

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No